CLINICAL TRIAL: NCT04456322
Title: A Randomized Non-inferiority Trial of Radiotherapy Plus Nimotuzumab or Cisplatin in Patients With Favorable Response to Induction Chemotherapy for Low-risk Locoregionally Advanced-Staged Nasopharyngeal Carcinoma
Brief Title: Radiotherapy Plus Nimotuzumab or Cisplatin in Nasopharyngeal Carcinoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Deputy Director of the Department of Nasopharyngeal Carcinoma, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-FXY-001
Record Dates: First submitted 2020-06-30; First posted 2020-07-02 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — nimotuzumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RT plus Nimotuzumab (Experimental): Patients with pretreatment plasma EBV DNA<1500 copy/ml and up to CR/PR according to RECIST and the EBV DNA reduced to undectable(0 copy/mL ) after two cycle induction chemotherapy ( TPF :Paclitaxel liposome135mg/m2 d1+DDP 25mg/m2 d1-d3+ 5-FU 750mg /m2/day civ120h, every 3 weeks for 2 courses) will have nimotuzumab (200mg, once a week during radiotherapy, a total of 7 weeks)
  Interventions: Drug: RT plus Nimotuzumab
- RT plus Cisplatin (Active Comparator): Patients with pretreatment plasma EBV DNA<1500 copy/ml and up to CR/PR according to RECIST and the EBV DNA reduced to undectable(0 copy/mL ) after two cycle induction chemotherapy( TPF :Paclitaxel liposome135mg/m2 d1+DDP 25mg/m2 d1-d3+ 5-FU 750mg /m2/day civ120h, every 3 weeks for 2 courses) will have concurrent cisplatin (100mg/m2, every three weeks,D1,D22,D43 of intensity modulated radiotherapy) )
  Interventions: Drug: RT plus Cisplatin

INTERVENTIONS:
Drug: RT plus Nimotuzumab — Nimotuzumab (200mg, once a week during radiotherapy, a total of 7 weeks)
  Arms: RT plus Nimotuzumab
Drug: RT plus Cisplatin — concurrent cisplatin (100mg/m2, every three weeks,D1,D22,D43 of intensity modulated radiotherapy )
  Other Names: Cisplatin
  Arms: RT plus Cisplatin

SUMMARY:
This is a phase III randomized clinical trial of definitive radiotherapy plus EGFR blocker nimotuzumab versus radiotherapy plus cisplatin(CCRT) for nasopharyngeal carcinoma (NPC) patients with favorable response to induction chemotheray(IC), determining whether radiotherapy combined with nimotuzumab was non-inferior to CCRT and may provide new evidence for individualized comprehensive treatment of locoregionally advanced NPC.

DETAILED DESCRIPTION:
Currently, NCCN (National Comprehensive Cancer Network) guidelines recommend induction chemotherapy combined with concurrent chemoradiotherapy as IIA level-evidenced treatment for locally advanced nasopharyngeal carcinoma (stage II-IVa). However, although induction chemotherapy combined with cisplatin based concurrent radiotherapy (CCRT) can significantly improve the survival of patients, the side effects during radiotherapy are more serious.

Previous studies have demonstrated that with a cut-off point of 1500 copies/mL, NPC patients could be segregated into a low-risk subgroup and a high-risk subgroup. Besides, our previous results showed that patients with plasma Epstein-Barr virus (EBV) DNA= 0 copy/mL and complete response/partial response (CR/PR) after induction chemotherapy had a significantly lower risk of disease progression than patients with plasma EBV DNA>0 copy/mL and stable disease /progressive disease (SD/PD),according to Response Evaluation Criteria in Solid Tumors (RECIST). As for these low-risk and chemotheray sensitive patients, it can be considered to reduce the current standard treatment intensity without affecting the survival rate of patients, which reduces the side effects of patients and improve the their life qualities.

Epidermal growth factor (EGFR) is an important therapeutic target for nasopharyngeal carcinoma. A retrospective study suggested that there was no significant difference in the 3-year overall survival between NPC patients who received nimotuzumab / cetuximab plus radiotherapy and those who received standard CCRT. Besides, in terms of hepatorenal toxicity, anti-EGFR drugs showed better safety compared with traditional cisplatin chemotherapy. Up to now, randomized clinical trial about the application of nimotuzumab after IC is still limited.

This is a phase III randomized clinical trial of definitive radiotherapy plus EGFR blocker nimotuzumab versus radiotherapy plus cisplatin for NPC patients with favorable response after IC, determining whether radiotherapy combined with nimotuzumab was non-inferior to CCRT after IC and may provide new evidence for individualized comprehensive treatment of locoregionally advanced NPC.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70, regardless of sex.
2. Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, type of WHO II or III, clinical stage II-IVa (except N3)(according to the 8th American Joint Committee on Cancer[AJCC] edition)
3. Patients with pre-treatment plasma EBV DNA<1500 copies/mL
4. Patients with plasma EBV DNA= 0 copy/mL and CR/PR according to RECIST after two cycle induction chemotherapy
5. ECOG (Eastern Cooperative Oncology Group) score: 0-1
6. Women in their reproductive years should ensure that they use contraception during the study period.
7. Hemoglobin (HGB) ≥90 g/L, white blood cell (WBC) ≥4×109 /L, platelet (PLT) ≥100×109 /L.
8. Liver function: Alanine transaminase(ALT), Aspartate aminotransferase(AST)< 2.5 times the upper limit of normal value (ULN), total bilirubin <2.0×ULN.
9. Renal function: serum creatinine <1.5×ULN
10. Patients must sign informed consent and be willing and able to comply with the requirements of visits, treatment, laboratory tests and other research requirements stipulated in the research schedule;

Exclusion Criteria:

1. Histologically confirmed keratinizing squamous cell carcinoma (WHO I)
2. Receiving radiotherapy or chemotherapy or targeted therapy previously
3. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
4. Suffered from other malignant tumors (except the cure of basal cell carcinoma or uterine cervical carcinoma in situ) previously.
5. Patients with significantly lower heart, liver, lung, kidney and bone marrow function.
6. Severe, uncontrolled medical conditions and infections.
7. At the same time using other test drugs or in other clinical trials.
8. Refusal or inability to sign informed consent to participate in the trial.
9. Other treatment contraindications.
10. Emotional disturbance or mental illness, no civil capacity or limited capacity for civil conduct.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2027-05-11 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years
  Defined from date of randomization to date of first documentation of progression or death due to any cause

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
  Defined from date of randomization to date of first documentation of death from any cause or censored at the date of the last follow-up.
Locoregional Relapse-Free Survival (LRFS) | 2 years
  Defined from date of randomization to date of first documentation of locoregional relapse or the date of death from any cause or until the date of the last follow-up visit
Distant Metastasis-Free Survival (DMFS) | 2 years
  Defined from date of randomization to date of first documentation of distant metastases or the date of death from any cause or until the date of the last follow-up visit
Objective Response Rate (ORR) | Three months after the completion of the CCRT with or without Nimotuzumab treatment
  An objective response is defined as either a confirmed CR or a PR, as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST1.1) from the National Cancer Institute (NCI)
Incidence rate of adverse events (AEs) | 2 years
  Analysis of acute and late adverse events (AEs) are evaluated. Numbers of patients of treatment-related adverse events(acute toxicity) as assessed by CTCAE v5.0.Numbers of patients of late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme.
Evaluate EGFR expression level and EGFR Gene Copy Number as a predictive marker for survival outcomes | 2 years
  Pre-treatment EGFR expression level and EGFR Gene Copy Number is evaluated by means of immunohistochemical testing and fluorescent in situ hybridization (FISH), respectively.
Change of QoL | 1 years
  QoL scores were assessed for each scale by using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTCQLQ-C30) before induction chemotherapy, before radiotherapy, at the end of radiotherapy, at 3 months after radiotherapy, at 6 months after radiotherapy and 12 months after radiotherapy
Change of EORTC quality of life questionnaire(QLQ) Head and Neck score | 1 years
  QoL scores were assessed by using EORTC quality of life questionnaire(QLQ) Head and Neck. The QLQ-H&N35 is composed of seven multi-item symptom scales (pain, swallowing, sensation, speech, eating from a social,perspective, social interactions, and sexuality) and 11 single-item symptom scales (teeth, opening mouth,dry mouth, sticky saliva,coughing, felt ill, pain medication use, nutritional supplementation, feeding tube requirement, weight loss, and weight gain). All of the scales and items ranged in score from 0 to 100. A high score for a functional or global QoL scale represents a relatively high/healthy level of functional or global QoL, whereas a high score for a symptom scale or item represents a high number of symptoms or problems.All of the scores mentioned above were assessed at the below time point:before induction chemotherapy, before radiotherapy, at the end of radiotherapy, at 3 months after radiotherapy, at 6 months after radiotherapy and 12 months after radiotherapy
Plasma EBV DNA copy number | 2 years
  Plasma EBV DNA copy number in both arms was assessed by Quantitative real time polymerase chain reaction(qRT-PCR) at pretreatment, after two cycle induction chemotherapy, during CCRT and follow up time . The predictive value of plasma EBV DNA copy number was assessed by survival analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Universitty Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Lee AW, Lau WH, Tung SY, Chua DT, Chappell R, Xu L, Siu L, Sze WM, Leung TW, Sham JS, Ngan RK, Law SC, Yau TK, Au JS, O'Sullivan B, Pang ES, O SK, Au GK, Lau JT; Hong Kong Nasopharyngeal Cancer Study Group. Preliminary results of a randomized study on therapeutic gain by concurrent chemotherapy for regionally-advanced nasopharyngeal carcinoma: NPC-9901 Trial by the Hong Kong Nasopharyngeal Cancer Study Group. J Clin Oncol. 2005 Oct 1;23(28):6966-75. doi: 10.1200/JCO.2004.00.7542. PMID 16192584
- [Background] Ribassin-Majed L, Marguet S, Lee AWM, Ng WT, Ma J, Chan ATC, Huang PY, Zhu G, Chua DTT, Chen Y, Mai HQ, Kwong DLW, Cheah SL, Moon J, Tung Y, Chi KH, Fountzilas G, Bourhis J, Pignon JP, Blanchard P. What Is the Best Treatment of Locally Advanced Nasopharyngeal Carcinoma? An Individual Patient Data Network Meta-Analysis. J Clin Oncol. 2017 Feb 10;35(5):498-505. doi: 10.1200/JCO.2016.67.4119. Epub 2016 Dec 5. PMID 27918720
- [Background] Blanchard P, Lee A, Marguet S, Leclercq J, Ng WT, Ma J, Chan AT, Huang PY, Benhamou E, Zhu G, Chua DT, Chen Y, Mai HQ, Kwong DL, Cheah SL, Moon J, Tung Y, Chi KH, Fountzilas G, Zhang L, Hui EP, Lu TX, Bourhis J, Pignon JP; MAC-NPC Collaborative Group. Chemotherapy and radiotherapy in nasopharyngeal carcinoma: an update of the MAC-NPC meta-analysis. Lancet Oncol. 2015 Jun;16(6):645-55. doi: 10.1016/S1470-2045(15)70126-9. Epub 2015 May 6. PMID 25957714
- [Background] Bossi P, Orlandi E, Bergamini C, Locati LD, Granata R, Mirabile A, Parolini D, Franceschini M, Fallai C, Olmi P, Quattrone P, Potepan P, Gloghini A, Miceli R, Mattana F, Scaramellini G, Licitra L. Docetaxel, cisplatin and 5-fluorouracil-based induction chemotherapy followed by intensity-modulated radiotherapy concurrent with cisplatin in locally advanced EBV-related nasopharyngeal cancer. Ann Oncol. 2011 Nov;22(11):2495-2500. doi: 10.1093/annonc/mdq783. Epub 2011 Mar 11. PMID 21398385
- [Background] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Background] Chan AT, Lo YM, Zee B, Chan LY, Ma BB, Leung SF, Mo F, Lai M, Ho S, Huang DP, Johnson PJ. Plasma Epstein-Barr virus DNA and residual disease after radiotherapy for undifferentiated nasopharyngeal carcinoma. J Natl Cancer Inst. 2002 Nov 6;94(21):1614-9. doi: 10.1093/jnci/94.21.1614. PMID 12419787
- [Background] Hou X, Zhao C, Guo Y, Han F, Lu LX, Wu SX, Li S, Huang PY, Huang H, Zhang L. Different clinical significance of pre- and post-treatment plasma Epstein-Barr virus DNA load in nasopharyngeal carcinoma treated with radiotherapy. Clin Oncol (R Coll Radiol). 2011 Mar;23(2):128-33. doi: 10.1016/j.clon.2010.09.001. Epub 2010 Oct 12. PMID 20943358
- [Background] Lin JC, Wang WY, Chen KY, Wei YH, Liang WM, Jan JS, Jiang RS. Quantification of plasma Epstein-Barr virus DNA in patients with advanced nasopharyngeal carcinoma. N Engl J Med. 2004 Jun 10;350(24):2461-70. doi: 10.1056/NEJMoa032260. PMID 15190138
- [Background] Liu LT, Tang LQ, Chen QY, Zhang L, Guo SS, Guo L, Mo HY, Zhao C, Guo X, Cao KJ, Qian CN, Zeng MS, Bei JX, Hong MH, Shao JY, Sun Y, Ma J, Mai HQ. The Prognostic Value of Plasma Epstein-Barr Viral DNA and Tumor Response to Neoadjuvant Chemotherapy in Advanced-Stage Nasopharyngeal Carcinoma. Int J Radiat Oncol Biol Phys. 2015 Nov 15;93(4):862-9. doi: 10.1016/j.ijrobp.2015.08.003. Epub 2015 Aug 7. PMID 26530755
- [Background] Huang CL, Sun ZQ, Guo R, Liu X, Mao YP, Peng H, Tian L, Lin AH, Li L, Shao JY, Sun Y, Ma J, Tang LL. Plasma Epstein-Barr Virus DNA Load After Induction Chemotherapy Predicts Outcome in Locoregionally Advanced Nasopharyngeal Carcinoma. Int J Radiat Oncol Biol Phys. 2019 Jun 1;104(2):355-361. doi: 10.1016/j.ijrobp.2019.01.007. Epub 2019 Jan 23. PMID 30682489
- [Background] Ciardiello F, Tortora G. A novel approach in the treatment of cancer: targeting the epidermal growth factor receptor. Clin Cancer Res. 2001 Oct;7(10):2958-70. PMID 11595683
- [Background] Mendelsohn J. Targeting the epidermal growth factor receptor for cancer therapy. J Clin Oncol. 2002 Sep 15;20(18 Suppl):1S-13S. No abstract available. PMID 12235219
- [Background] Ramakrishnan MS, Eswaraiah A, Crombet T, Piedra P, Saurez G, Iyer H, Arvind AS. Nimotuzumab, a promising therapeutic monoclonal for treatment of tumors of epithelial origin. MAbs. 2009 Jan-Feb;1(1):41-8. doi: 10.4161/mabs.1.1.7509. PMID 20046573
- [Background] You R, Sun R, Hua YJ, Li CF, Li JB, Zou X, Yang Q, Liu YP, Zhang YN, Yu T, Cao JY, Zhang MX, Jiang R, Mo HY, Guo L, Cao KJ, Lin AH, Qian CN, Sun Y, Ma J, Chen MY. Cetuximab or nimotuzumab plus intensity-modulated radiotherapy versus cisplatin plus intensity-modulated radiotherapy for stage II-IVb nasopharyngeal carcinoma. Int J Cancer. 2017 Sep 15;141(6):1265-1276. doi: 10.1002/ijc.30819. Epub 2017 Jun 23. PMID 28577306
- [Background] Lin M, You R, Liu YP, Zhang YN, Zhang HJ, Zou X, Yang Q, Li CF, Hua YJ, Yu T, Cao JY, Li JB, Mo HY, Guo L, Lin AH, Sun Y, Qian CN, Ma J, Mai HQ, Chen MY. Beneficial effects of anti-EGFR agents, Cetuximab or Nimotuzumab, in combination with concurrent chemoradiotherapy in advanced nasopharyngeal carcinoma. Oral Oncol. 2018 May;80:1-8. doi: 10.1016/j.oraloncology.2018.03.002. Epub 2018 Mar 13. PMID 29706183